CLINICAL TRIAL: NCT05763524
Title: European Multicenter Study on Role of Lymph Node Dissection in Surgical Management of Adrenal Cortical Carcinoma
Acronym: LACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5171
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; Lymphadenectomy; Eurocrine
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Adrenalectomy; Lymph Node Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenalectomy in patients operated for Adrenocortical Carcinoma: All adult (18 years old and older) patients registered in EUROCRINE® database that underwent surgery for adrenocortical carcinoma from 2015 till 2021 will be included
  Interventions: Procedure: Adrenalectomy with or without lymphadenectomy

INTERVENTIONS:
Procedure: Adrenalectomy with or without lymphadenectomy — Regarding lymphadenectomy extent, it will be described as locoregional or systematic depending on availability of data in the Eurocrine database.

SUMMARY:
This project will evaluate of the number of patients who underwent adrenalectomy for ACC in different European centers using the EUROCRINE® database. The analysis will focus on the extent of lymph nodal dissection (i.e. number of lymph nodes and nodal stations dissected during adrenalectomy). We aim to evaluate the oncologic radicality of surgical treatment and the rate of tumour recurrences after surgery and nodal metastasis related to the stage of the disease and to tumour side (left/right).

DETAILED DESCRIPTION:
Adrenocortical carcinoma (ACC) is a rare malignancy with an estimated annual incidence of only 0.5 to 2.0 per million population and a high rate of mortality: Stage I, II and III 5 years-survival is respectively 84%, 63% and 24%, while medium survival is less than 12 months for metastatic disease. Stage of the disease, age at diagnosis, tumour grading and complete surgical resection are the main prognostic factors. Surgical treatment is the only effective therapeutic strategy for ACC and recent guidelines recommend loco-regional lymph node dissection as a fundamental surgical element in order to guarantee complete resection. However, adrenal lymphatic drainage can be variable. The main collecting lymph nodes representing the first tiers in the lymphatic drainage are the peri-adrenal nodes and the renal ilum nodes. In addition, the posterior lymphatic drainage flows to lymph nodes located posterior to the IVC, and on the right edge of the aorta for the right adrenal gland, or on its right left edge for the left gland, stretching from the celiac region near the diaphragmatic crus to the renal vessels.

The anterior lymphatic drainage flows downward to the lumboaortic nodes and ends in the interaortocaval space, on the right edge of the aorta for the right adrenal gland, and on its right left edge for the left gland and mainly around the renal hilum. Collecting nodes can be located below the renal pedicle, sometimes extending as far as the origin of the iliac vessel. Most authors concur in describing a lymphatic drainage that passes through the diaphragm directly into the posterior mediastinal nodes. A majority of lymphatic channels run medially to the thoracic duct, often without the involvement of any lymph nodes. Furthermore, it is impossible to predict which pathway would be involved in case of a malignant lesion, because all pathways would probably be involved simultaneously because of the size, often >10 cm, of ACC at diagnosis, and considering that the lymphatic stream can be disorganized because of the tumour volume or lymph node involvement. Therefore, the extent of lymph node dissection in order to involve other stations should be considered only on the basis of pre-operative radiological evidence and intra-operative evaluation. Despite aggressive surgical resection, local and distant recurrence rate after R0 surgery remains as high as 50-80%, potentially because of the lack of an accurate identification of the nodes stations for the lymph node dissection. Indeed, nodes drain disorganization due to the high tumour volume makes impossible to predict accurately the lymphatic metastatic pathway. In this context, the rarity of ACC leads to heterogeneity of the scientific studies and consequently to the lack of perspective works, so that tumour recurrence evaluation refers to patients categories who underwent lymph node dissection with or without preoperative evidence of nodal disease

ELIGIBILITY:
Inclusion Criteria: All adult (18 years old and older) patients that underwent surgery with a final histology of adrenocortical carcinoma from 2015 till 2021

Inclusion Criteria:

* All adult (18 years old and older) patients
* underwent surgery
* final histology of adrenocortical carcinoma
* among European centers that participate in the Eurocrine® database between 2015 and 2021

Exclusion Criteria:

* Patients <18 years old
* Patients with metastatic disease at time of clinical referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with final histology of adrenocortical carcinoma operated among European centers that participate in the Eurocrine® database between 2015 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adrenocortical Carcinoma (ACC) among European endocrine centers | January 2015- January 2021
  Identification of the number of patients who underwent adrenalectomy for diagnosis of ACC among European centers participating in the Eurocrine database
Extent of lymphadenectomy | January 2015- January 2021
  Evaluation of the lymph node dissection extension (in terms of number of lymph nodes and nodal stations dissected during surgical treatment for ACC)

SECONDARY OUTCOMES:
Oncologic outcomes | January 2015- January 2021
  Descriptive analysis of oncologic outcome (in terms of disease recurrence, lymph node metastasis and their association to the tumour stage) in patients who underwent surgical treatment of ACC in European centers

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Prof, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests will be evaluated by the Eurocrine Council